CLINICAL TRIAL: NCT02460510
Title: Role of Hypertonic Saline Versus Mannitol in the Management of Raised Intracranial Pressure in Patients With ALF: A Randomized Open -Label Study
Brief Title: Role of Hypertonic Saline Versus Mannitol in the Management of Raised Intracranial Pressure in Patients With ALF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ALF-01
Record Dates: First submitted 2015-05-25; First posted 2015-06-02 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Acute Liver Failure
MeSH Terms: conditions — Liver Failure, Acute | interventions — Mannitol; Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mannitol (Experimental): Treatment with mannitol intravenous (IV) bolus over 20 to 30 minutes. The dose is 0.25 g/kg IV as a 20% solution repeated every 4th hourly.(8) Mannitol infusion to be stopped if s osmolarity >320mm
  Interventions: Drug: Mannitol
- 3% hypertonic saline (Active Comparator): Treatment with 3% hypertonic saline as continuous infusion. Continuous 3% NaCl infusion to be started at a rate of 25ml /hr and titrated q4hrs per sliding scale to achieve a target serum sodium level of <160 mmol/L.
  Interventions: Drug: 3% hypertonic saline

INTERVENTIONS:
Drug: Mannitol
  Arms: Mannitol
Drug: 3% hypertonic saline
  Arms: 3% hypertonic saline

SUMMARY:
Patients with ALF (Acute liver Failure) would undergo a detailed clinical evaluation. Information would be collected regarding the onset and duration of symptoms, etiology, and severity of disease, other baseline clinical features, demographic characteristics, routine biochemical and hematological investigations. Patients would also be screened for the assessment of raised intracranial hypertension by either clinical or neuroimaging or by ONSD (optic nerve sheath diameter) and TCD (Transcranial doppler ultrasonography). Patient found to be having risen ICP (Intra Cranial Pressure) would be randomized in the two groups of the study. The group A would receive intravenous mannitol 20 to 30 minutes every 4 hourly where as those in the group B would be given 3% hypertonic saline as continuous infusion at a rate of 25ml /hr and titrated q4 hrs per sliding scale to achieve a target serum sodium level of 144-155 mmol/L .Both the groups would receive other supportive measures such as head end elevation, oxygen supplementation, dextrose infusion to maintain normoglycemia standard medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Acute Liver Failure with age >18 yrs
* Grade III or grade IV HE with raised ICP
* Patient's next-of-kin consenting for the study protocol.

Exclusion Criteria:

* Patients with ocular trauma.
* K/c/o DCM, congestive heart failure, cerebral aneurysm, intracranial pathology
* Serum Na>160 and s creat>1.5 mg% with oligurea

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
To study response to therapy at 12 hr in HTS Vs mannitol group in reduction of ICP (Intra Cranial Pressure) | 12 hours
  ICP (Intra Cranial Pressure) as assessed by ONSD (Optic Nerve Sheet Diameter) < 5mm PS<1.2 Pupils - RTL(reaction to light) {if initially NTR(no reaction to light)} BP<150/90(if initially high) Pulse >60( if < 60)

SECONDARY OUTCOMES:
Correlation of arterial NH3 to raised ICT (Intra cranial Tension). | 2 years
Survival. | 28 days
Length of ICU/hospital stay. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India